CLINICAL TRIAL: NCT01823497
Title: Parent/Nurse Controlled Analgesia for Post-Operative Pain Management in Neonates: A Preliminary Randomized Controlled Trial
Brief Title: Parent/Nurse Controlled Analgesia in the Neonatal Intensive Care Unit
Acronym: PNCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP4155
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Abdominal Surgery; Thoracic Surgery
Keywords: Neonatal Intensive Care Unit; neonate; pain; morphine; Parent/Nurse Controlled Analgesia
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent/Nurse Controlled Analgesia (Active Comparator): Parent/Nurse Controlled Analgesia will be the method of morphine delivery.
  Interventions: Drug: Morphine
- Continuous Opioid Infusion (Active Comparator): Continuous Opioid Infusion will be the method used to deliver morphine to group 2
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Morphine will be used to control pain post-surgery.

SUMMARY:
The aim of this study is to examine the safety and effectiveness of 2 morphine delivery systems for post-surgical neonates. The investigators hypothesize that this study will be feasible to conduct, and that neonates receiving morphine via a Parent/Nurse Controlled Analgesia pump will receive less morphine and experience fewer side effects than neonates receiving morphine via continuous opioid infusion.

ELIGIBILITY:
Inclusion Criteria:

* Surgery Location:

  * Abdominal or Thoracic
  * First surgery only

Age:

* Born ≥ 34-44 weeks post-menstrual age
* Weight: Weight at birth or current weight ≥2 kg Intubated or extubated

Prior opioid exposure:

* < 2 days of continuous exposure
* if history of > 2 day continuous exposure, must be off continuous drip for a week
* Intermittent exposure ≤ 2 days prior to surgery Neonates exposed to chronic opioids in utero *In utero exposure to Selective Seretonin Reuptake Inhibitors and illicit drugs will be screened for and annotated.

At least 1 parent is English-speaking

Exclusion Criteria:

* Surgery Type:

  * Cardiac, Patent Ductus Arteriosus Ligation; Omphalocele (if intubated pre-operatively)

Diagnoses:

• Necrotizing Enterocolitis; Diaphragmatic hernia (unless thoracoscopically repaired); Chemically or physiologically paralyzed Receiving vasopressors Receiving acetaminophen or a benzodiazepine (lorazepam or midazolam) ≤ 24 h before surgery Patients with any of the following: Epidural; Oscillating ventilator

Ages: 1 Minute to 70 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keri R Hainsworth, PhD, Principal Investigator — Medical College of Wisconsin; Michelle L Czarnecki, MSN RN-BC CPNP, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parent/Nurse Controlled Analgesia | Continuous Opioid Infusion
Started | 19 | 17
Completed | 16 | 9
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent/Nurse Controlled Analgesia | Continuous Opioid Infusion | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 9 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 4 [1.3 to 12.0] | 2 [0.0 to 59.0] | 4 [2.0 to 11.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 14 | 9 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 14 | 2 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption
Description: The investigators will measure amount of morphine consumed post-surgery in mg/kg/hour
Time Frame: 5 days post surgery
Measure: Median (Inter-Quartile Range); unit: mg/kg/hr
Arm/Group | Parent/Nurse Controlled Analgesia | Continuous Opioid Infusion
Number analyzed (Participants) | 16 | 9
mg/kg/hr | 0.014 [0.013 to 0.017] | 0.036 [0.036 to 0.040]

2. Secondary Outcome: Revised-Face, Legs, Activity, Cry, Consolability (Revised-FLACC) Scale
Description: The investigators will report the average pain score per POD, for 4 days (PODs 0,1,2,3). Higher scores mean worse outcome. Good pain control will be defined as pain less than 4 on a 0-10 scale. Pain is scored by observers on a minimum of 0 (no pain) to a maximum of 10 (worst pain) on this scale. The median and inter-quartile range of the average pain score per post-operative day is reported. The timeframe includes the post-operative day (POD 0), and 3 days post-surgery (POD 1-3), for a total of 4 post-operative days.
Time Frame: 4 days post surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Parent/Nurse Controlled Analgesia | Continuous Opioid Infusion
Number analyzed (Participants) | 16 | 9
units on a scale
  Post-operative Day 0 | 1.25 [0.43 to 2.81] | 1.67 [0.00 to 4.42]
  Post-operative Day 1 | 1.79 [1.37 to 2.55] | 1.083 [0.00 to 3.18]
  Post-operative Day 2 | 2.17 [0.31 to 2.36] | 1.83 [0.58 to 3.42]
  Post-operative Day 3 | 1.00 [0.00 to 2.44] | 1.25 [0.31 to 2.45]

3. Other Pre Specified Outcome: Methadone Use
Description: Methadone will serve as a surrogate for tolerance and will be monitored up to 3 days after the morphine has been discontinued.
Time Frame: up to 3 days after morphine is discontinued
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 3 post-operative days
Description: The intervention involved in this study would not be associated with all-cause mortality
Arm/Group | Parent/Nurse Controlled Analgesia | Continuous Opioid Infusion
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 7/16 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parent/Nurse Controlled Analgesia (N=16) | Continuous Opioid Infusion (N=9)
Naloxone, reintubation, or methadone (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Sedation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT01823497/Prot_SAP_000.pdf